CLINICAL TRIAL: NCT00481130
Title: Alport Syndrome Treatments and Outcomes Registry
Acronym: ASTOR
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0704M05941
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alport Syndrome
Keywords: Alport Syndrome; x linked; autosomal dominant Alport syndrome; glomerular basement membrane; hereditary nephritis; familial benign haematuria; type IV collagen; hereditary nephritis with neurosensory deafness; vison loss
MeSH Terms: conditions — Nephritis, Hereditary; Alport syndrome, dominant type

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
ASTOR's primary purpose is to enroll families and patients with a history of Alport syndrome in a central registry. The information we gather will be used as a basis for studies designed to test potential treatments for Alport syndrome. ASTOR also aims to provide patients, families and physicians with the most up-to-date information about Alport syndrome.

DETAILED DESCRIPTION:
The University of Minnesota's Department of Pediatrics has created the Alport Syndrome Treatments and Outcomes Registry (ASTOR). ASTOR's primary purpose is to enroll families and patients with a history of Alport syndrome in a central registry. The information we gather will be used as a basis for studies designed to test potential treatments for Alport syndrome. ASTOR also aims to provide patients, families and physicians with the most up-to-date information about Alport syndrome.

You can help doctors learn more about Alport syndrome and test possible treatments for the disease by enrolling in ASTOR. Since Alport syndrome is a rare disease it is essential for ASTOR to enroll as many patients as possible. Together, you and others facing the challenges of Alport syndrome can provide valuable information that will help doctors better understand the disease and in turn, help patients with Alport syndrome now and in the future.

ELIGIBILITY:
Inclusion Criteria: History of a diagnosis of Alport syndrome, Family or individuals need to be able to comprehend the consent and HIPAA forms written in the English language.

Exclusion Criteria: Uncertain diagnosis of Alport syndrome.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family and individual history of a diagnosis of Alport syndrome
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2007-09; Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Data Collection: natural history study | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Kashtan, MD, Principal Investigator — University of Minnesota, Department of Pediatrics
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kashtan CE, Gross O. Clinical practice recommendations for the diagnosis and management of Alport syndrome in children, adolescents, and young adults-an update for 2020. Pediatr Nephrol. 2021 Mar;36(3):711-719. doi: 10.1007/s00467-020-04819-6. Epub 2020 Nov 6. PMID 33159213